CLINICAL TRIAL: NCT04060173
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1b Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ABP-671 Administered Orally for 10 Days in Subjects With Hyperuricemia
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ABP-671
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABP-671-102
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Hyperuricemia; Gout
Keywords: Gout; Hyperuricemia
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with ABP-671 (Experimental): Three sequential dose escalation cohorts of ABP-671 administered orally for 10 days.
  Interventions: Drug: ABP-671
- Treatment with placebo (Placebo Comparator): Three sequential dose escalation cohorts of ABP-671 matching placebo administered orally for 10 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ABP-671 — ABP-671 is an investigational drug
  Arms: Treatment with ABP-671
Other: Placebo — Matching placebo
  Arms: Treatment with placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of ABP-671 administered orally in subjects with hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be medically documented as healthy and acceptable at screening.
* Subjects must have serum uric acid level at screening ≥ 7.0 mg/dL for men, ≥ 6.0 mg/dL for women.
* Subjects must have a Body Mass Index (BMI) between 18.0 and 34.0 kg/m2 (inclusive).
* Subjects must have a body weight of 50 kg or higher.
* The subject agrees to abstain from alcohol consumption for 48 hours prior to dosing, for the duration of the in-house study period, and for 48 hours prior to each in-clinic follow up visit.
* The subject is a nonsmoker.
* Women must be non-pregnant and non-lactating, and either surgically sterile or postmenopausal for ≥ 12 months.
* Men must be surgically sterile, abstinent or if engaged in sexual relations with a female partner of child-bearing potential, the participant must be using a condom with spermicide from Screening and for a period of 30 days after the last dose of Study Drug. The Investigator will assess the adequacy of methods of contraception on a case-by-case basis.
* Subjects must have a complete blood count (CBC) and platelet count within the normal range or considered not clinically significant by the principal investigator.
* Other than elevated serum uric acid, subjects must have normal blood chemistry or results considered not clinically significant by the investigator.
* Subjects must have a normal urinalysis or results considered not clinically significant by the investigator including a normal protein/creatinine ratio per local lab reference ranges (≤ 200 mg/g) and a urine creatinine result that does not exceed 300 mg/dL. Any out of range values may be repeated per Investigator discretion.
* Subjects must have a normal ECG or results considered not clinically significant by the principal investigator.
* Subjects must be able to comply with the study and follow-up procedures.
* Subjects are able to understand the study procedures and risks involved and must provide signed informed consent to participate in the study.

Exclusion Criteria:

* Subjects with any history or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urological, or psychiatric disorders.
* Subjects who are positive for human immunodeficiency virus (HIV), Hepatitis B surface antigen, and/or Hepatitis C virus.
* Subjects who have used prescription drugs, over-the-counter drugs, or herbal remedies within 3 weeks before Day 1 of study medication dosing.
* Subjects who are positive for urine drug and alcohol screening tests.
* Subjects who have undergone major surgery within 3 months prior to Day 1.
* Women who are pregnant or breastfeeding.
* Subjects who received any investigational test article within 5 half-lives or 30 days, whichever is longer, prior to Day 1 study medication dosing.
* Recent blood donation for more than 500 mL within 2 months of screening.
* Abnormal ECG including QTc > 470 (F) and > 450 (M).
* Subjects who consumed Seville oranges- or grapefruit-containing foods or beverages within 7 days before Day 1 and during the entire study duration.
* Subjects with any condition that, in the judgment of the investigator, would place him/her at undue risk, or potentially compromise the results or interpretation of the study.
* Prior exposure to ABP-671.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 38 days
  Measured by the number of patients with AEs

SECONDARY OUTCOMES:
Maximum observed plasma concentration of ABP-671 (Cmax) | 2 weeks
Area under time-concentration curve (AUC) | 2 weeks
Time of maximum observed plasma concentration of ABP-671 (Tmax) | 2 weeks
Volume of distribution (Vd) | 2 weeks
Half life of ABP-671 (t1/2) | 2 weeks
The effect of ABP-671 versus placebo on the percent change from baseline in serum uric acid | 24 days
The effect of ABP-671 versus placebo on change in urine uric acid excretion | 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States